CLINICAL TRIAL: NCT02996903
Title: Prospective Multicenter Registry On RadiaTion Dose Estimates Of Cardiac CT AngIOgraphy IN Daily Practice in 2017
Acronym: PROTECTION-VI
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Thomas Stocker, Co-Principal Investigator, LMU Klinikum
Other Study IDs: MUC I002-16
Record Dates: First submitted 2016-12-13; First posted 2016-12-19 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Cardiac Disease; Malignancy, Second
Keywords: Cardiac Computed Tomography (CT) Angiography (CCTA); coronary artery disease; malignancy induction; radiation dose; dose saving techniques; effective dose
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The "Prospective Multicenter Registry On RadiaTion Dose Estimates Of Cardiac CT AngIOgraphy IN Daily Practice in 2017" (PROTECTION-VI) study is a prospective registry and investigator-initiated initiative without third-party funding, which will collect and analyze the radiation dose exposure of Cardiac Computed Tomography Angiographic (CCTA) studies in current daily practice worldwide. Particularly, the study will assess the use of strategies for dose reduction during CCTA.

A decade ago, the multicentre observational PROTECTION-I study has revealed that the dose-length-product of CCTA ranges between 568 - 1259 mGy x cm with a median of 885 mGy x cm. This corresponds to an estimated effective dose of approximately 12 mSv. Since then a variety of techniques have been developed and enhanced in order to reduce radiation exposure during CCTA. Recent studies demonstrated feasibility of dramatically reduced effective radiation doses during CCTA (0,1 - 0,3 mSv). This has been executed in small cohorts of patients at scientific expert centers. However, it remains unclear, if such low-level radiation dose exposure may be achieved in clinical routine and if diagnostic image quality is maintained. In order to analyze the magnitude of radiation dose exposure of CCTA in today's clinical practice and the current use of dose-saving techniques, we designed the PROTECTION-VI study. Eventually, this study may contribute to further improving radiation dose exposure for patients undergoing CCTA.

DETAILED DESCRIPTION:
Cardiac CT angiography (CCTA) has emerged to a powerful and commonly used diagnostic tool for the evaluation of coronary artery disease. Advantages of CCTA are its non-invasive approach, widespread availability and high negative predictive value to rule out coronary artery disease. However, radiation exposure during CCTA needs to be considered, due to the potential risk of malignancy induction.

A decade ago, the multicentre observational PROTECTION I study has revealed that the dose-length-product of CCTA ranges between 568-1259 mGy x cm with a median of 885 mGy x cm. This corresponds to an estimated effective dose of approximately 12 mSv. Furthermore, PROTECTION I demonstrated an up to 7-fold variation of radiation dose between different study sites implicating the large potential for dose reduction. Finally, significant differences have been detected in the radiation exposures between CT systems from different vendors and application of dose-saving algorithms, implying that approaches for dose reduction with respect to hardware and software have also been of relevance in 2007.

Since then a variety of techniques have been developed and enhanced in order to reduce radiation exposure during CCTA. Earlier, ECG-controlled tube current modulation has been accepted to reduce radiation dose and was therefore used in ECG-gated retrospective cardiac spiral scanning.

Another dose-saving technique is the reduction of tube potential from conventionally 120 kVp to 100 kVp in non-obese patients. In the PROTECTION II trial we demonstrated that diagnostic image quality is being maintained with a reduction of tube potential to 100 kVp while radiation exposure was significantly reduced by 31%.

Development of prospective ECG-gated axial (sequential) scanning allowed further dose reduction, due to administration of radiation only at the end of diastole. In the PROTECTION III trial we could demonstrate that diagnostic image quality is being maintained with prospective ECG-gated axial scanning in patients with stable and low heart rates while radiation exposure was reduced by 69% when compared to conventional spiral scanning with retrospective ECG gating. Using prospectively ECG-triggered high-pitch spiral CCTA with image acquisition during only one cardiac cycle, additional dosage may be saved when used in selected patients with low and stable heart rates. However, a scan strategy with an attempt of high-pitch scanning first is vulnerable to motion artefacts and bears the risk of repeated scanning.

In the PROTECTION IV trial we compared a scan strategy of high-pitch helical scanning first with a conventional scan first strategy. We could demonstrate maintenance of image quality using the strategy of high-pitch helical scanning first, while radiation exposure was reduced by 57 %, when compared to the conventional scan first strategy.

The introduction of iterative image reconstruction technique with advanced raw data processing let to improvement of image quality compared to traditional filtered back projection. This allowed additional dose saving during image acquisition. In the PROTECTION V trial we demonstrated the feasibility of combining iterative image reconstruction techniques with a reduction of tube currents by 30% leading to maintenance of diagnostic image quality while saving radiation dose linearly to tube current.

In summary, the four randomized clinical trials PROTECTION II-V demonstrated that different techniques for reducing radiation exposure during CCTA can be applied in clinical practice without compromising diagnostic image quality. The studies show that the different approaches can also be applied in combination and that these approaches can be used with different CT platforms from different CT vendors.

Recent studies demonstrated that the effective radiation dose for one CCTA scan may be reduced to 0,3 mSv15 or even below 0,1 mSv in a small amount of carefully selected patients. However, it remains unclear if such dramatically low dosages are being achieved and if diagnostic image quality is being maintained in clinical routine. In order to analyze the magnitude of radiation dose exposure during CCTA in today's clinical practice, we designed the international and multicentric PROTECTION VI study. We will assess the variation of radiation dose with respect to vendors, CT systems and study sites. Furthermore, we will evaluate the usage of dose saving strategies including the above-mentioned in daily practice and analyze their effect on diagnostic image quality. On the basis of the collected data, we will evaluate the potential use of additional dose savings for each site individually.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical indication for CCTA in order to evaluate the coronary arteries or other cardiac structures
* Patients age > 18 years
* Signed informed consent (if required by local IRB)

Exclusion Criteria:

* Known allergy to contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Cardiac Computed Tomography Angiography (CCTA) in clinical routine.
Sampling Method: Probability Sample
Enrollment: 4502 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Radiation dose estimates of cardiac CT angiographies in daily practice | Baseline
  Assessment after CT scan by radiologist or technical assistant, documented on questionnaire.

SECONDARY OUTCOMES:
Use of dose-saving strategies | Baseline
  Use of Low tube potential imaging, Low tube current imaging, Automated Exposure Control, ECG-controlled tube current modulation (dose pulsing), Iterative image reconstruction techniques and Scan protocols (Prospective ECG-triggered axial scanning technique, Prospective ECG-triggered high-pitch spiral acquisition) will be assessed in the Core Lab according to information given by the CT-examiner on a questionnaire.
Assessment of CCTA image quality in relation to radiation dose | Baseline
  Assessment after CT scan by CT-examiner on questionnaire (qualitative) or in the Core Lab (quantitative).
  Quantitative Assessment includes Signal intensity, Image noise, Contrast-to-noise ratio, Signal-to-noise ratio. Qualitative assessment of each coronary artery is performed using a 3-point grading scale including excellent, intermediate or non-diagnostic as documented on a provided questionnaire.
Sufficient result of the first CCTA scan or need for repeated scans | Baseline
  According to information given by the CT-examiner on a questionnaire.
Cardiac CT scan length and relationship between scan and heart length | Baseline
  Assessment in Core Lab after analysis of CT scans.
Comparison of dose estimates between different continents, CT vendors and CT systems | Baseline
  Analysis done in the Core Lab according to information given by the CT-examiner on a questionnaire.

CONTACTS AND LOCATIONS:
Locations (4):
- National Heart, Lung, and Blood Institute, Bethesda, Maryland, United States
- University of British Columbia, Department of Medical Imaging, Vancouver, British Columbia, Canada
- Ludwig-Maximilians-Universitaet Muenchen, Medizinische Klinik I, Munich, Bavaria, Germany
- Technion Israel Institute of Technology, The Ruth and Bruce Rappaport Faculty of Medicine, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stocker TJ, Leipsic J, Hadamitzky M, Chen MY, Rubinshtein R, Deseive S, Heckner M, Bax JJ, Kitagawa K, Marques H, Schmermund A, Silva C, Mahmarian J, Kang JW, Grove EL, Lesser J, Massberg S, Hausleiter J. Application of Low Tube Potentials in CCTA: Results From the PROTECTION VI Study. JACC Cardiovasc Imaging. 2020 Feb;13(2 Pt 1):425-434. doi: 10.1016/j.jcmg.2019.03.030. Epub 2019 Jun 12. PMID 31202772